CLINICAL TRIAL: NCT04790760
Title: Glucose Differences Between the Left Arm and Right Arm in Diabetic Patients Using a Continuous Glucose Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Pacific (Other)
Collaborators: Manshadi Heart Institute, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-29
Record Dates: First submitted 2021-02-19; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continuous Glucose Monitoring (Experimental): Participants will wear a CGM device on the back of both their left and right arm for 6 weeks.
  Interventions: Dietary Supplement: Supplement Consumption; Device: Continuous Glucose Monitors

INTERVENTIONS:
Dietary Supplement: Supplement Consumption — Participants will consume one 500 mg cinnamon capsule and one 300 mg aloe vera capsule twice per day for weeks 3-6.
Device: Continuous Glucose Monitors — Participants will wear a CGM on the back of their left and right arm for weeks 1-6.

SUMMARY:
Continuous glucose monitoring (CGM) is an emerging field for diabetes management. CGMs are small devices primarily placed on a patient's upper arm that allow providers and patients to individualize therapy by looking at real time glucose levels. While the accuracy of these devices is extensively researched, there are no large-scale studies evaluating the differences between left and right arm glucose readings in the diabetic population. Additionally cinnamon and aloe vera are supplements commonly used by diabetic patients to help improve glycemic control. However, there remains a shortage of studies researching the effects of cinnamon and aloe vera on diabetic patients' glycemic control.

The purpose of this study is to determine if there is a difference between glucose levels in the right arm and left arm in diabetic patients and to evaluate if cinnamon and aloe vera supplements impact glycemic control in diabetic patients.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) is an emerging field for diabetes management. CGMs allow providers to individualize therapy by looking at real time glucose levels, detect changes in glucose and raise awareness for hypo- and hyperglycemic events.[1] Some CGMs can be placed on the patient's arm to monitor glucose at regular intervals. The data is downloaded onto a reader where it can be viewed or sent to a computer for more in depth analysis. There are multiple Food and Drug Administration (FDA) approved CGM devices. The FDA considers a device to be accurate if 99% of glucose measurements are within 20% of lab results and if 95% of glucose measurements are within 15% of lab results.[2]

The accuracy and precision of CGMs is improving with increased use and advancement of the systems in use. CGM data has been deemed accurate for self use to adjust insulin dosage, detection of hypoglycemia and determining the clinical response to therapy.[3] However, CGMs are a new technology and while they have vastly improved since they originally came to market, there are still many concerns over their accuracy and ability to inform clinical treatment decisions.[3] An analysis conducted on the reports to the FDA Manufacturer and User Facility Device Experience (MAUDE) database since 2015 revealed over 25,000 complaints of CGM inaccuracy.[4]

In the American Diabetes Association (ADA) 2020 Guidelines on the Standards of Medical Care in Diabetes, it is stated that glycemic goals are achieved through glucose monitoring and, as such, self monitoring blood glucose is essential for reaching these goals.[5] CGMs are used to guide the treatment of diabetes including pharmacologic intervention, recommendations for hypoglycemia prevention and nutrition goals. The recommended time spent in range, time above range and time below range are also outlined in these guidelines.[5] The significance of time below range is associated with the risk of hypoglycemia. The more time spent below range is going to increase the chance of experiencing a hypoglycemic event which, if experienced, will have both negative physical and psychological effects on the person. In the most severe cases it can also lead to seizures, coma and death.[5] Increased time spent above range has been directly correlated with incidence and progression of microvascular complications associated with diabetes like retinopathy, neuropathy and kidney disease.[5] Time spent in range is also significant because in addition to informing treatment decisions, it has also been correlated to improvements in hemoglobin A1c (HbA1c). In a recent analysis of 18 studies reporting paired HbA1c and time in range (%), it was found that for every 10% change in time in range, there was a corresponding 0.8% change in HbA1c.[6] This could mean that if a person spends 10% more time in range, their HbA1c may reduce up to 0.8%. This is significant since HbA1c is a gold standard marker of glycemic control in the diabetic population.[5]

Based on previous studies, the evaluation of CGM readings in the left and right arms of diabetic patients is needed. The information provided by CGMs outside of glucose levels such as time range information, hyper- or hypoglycemic glucose levels, and even immediate phone alerts for very low or very high readings in newer devices highlights the ever growing and critical role these devices play in the care of diabetic patients, and as such their accuracy and proper use is of the utmost importance.[7]

Cinnamon and aloe vera supplements are available over the counter and are used by consumers for many different ailments. Both cinnamon and aloe vera have been used for several centuries across many different cultures for a wide range of medicinal purposes. Diabetes is an example of one of the disease states commonly targeted by these two supplements. Patients with diabetes frequently consume cinnamon and aloe vera dietary supplements in an effort to improve their glycemic control. As research into the effects of these supplements has expanded, the understanding of their safety and practical uses has become better understood and is generally accepted.[8,9] There are many dietary supplements or food classified cinnamon and aloe vera based products on the market. Both cinnamon and aloe vera are Generally Recognized As Safe (GRAS status). However there is a lack of long term evaluation of the effects of these supplements in the diabetic patient population.

This study is a controlled, prospective trial that aims to evaluate the difference in glucose readings between the right arm and left arm using continuous glucose monitors in diabetic patients. In addition this study aims to evaluate the effect of cinnamon and aloe vera supplementation on glycemic control in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-65 years of age
* Diagnosed with type 2 diabetes
* Willing to wear CGM for 6 weeks on both arms
* Willing to come in for 4 office visits over 6 weeks
* Willing to consume assigned supplement twice a day for 4 weeks
* Willing to receive and respond to daily text messages or maintain a daily study log of supplement consumption
* Have active health insurance
* Willing to refrain from any heat therapy for the duration of the study
* Willing to refrain from taking any other supplements that are deemed by the investigator to alter glucose for the duration of the study
* Willing to refrain from consuming ascorbic acid and salicylic acid for the duration of the study due to a known interaction with CGMs
* Be able to self-monitor blood glucose with finger-stick method
* Have a baseline HbA1c > 6.5%

Exclusion Criteria:

* Any active dermatologic condition on the upper arms
* Implanted medical devices (i.e. pacemaker)
* Critically ill or dialysis patients
* Planned magnetic resonance imaging screening, computed tomography scan, x-ray imaging or high-frequency electrical heat treatment during study period
* Current systemic infections
* Participants who are unable to fully understand the study or consent process will not be included in the study due to the lack of a qualified medical translator
* Change in diabetic medication regimen within the previous 30 days (except insulin)
* Self-identified allergy to cinnamon or aloe vera
* Refusal to sign the informed consent document
* Pregnant, planned-pregnancy during study period or currently breast-feeding
* History of hypoglycemic episodes warranting medical attention experienced in the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Difference in time-matched glucose levels between the right arm and the left arm | 6 weeks

SECONDARY OUTCOMES:
Difference in time in range between the right arm and the left arm | 6 weeks
Difference in time above range between the right arm and the left arm | 6 weeks
Difference in time below range between the right arm and the left arm | 6 weeks

OTHER OUTCOMES:
Change in continuous glucose monitor measured glucose levels | 6 weeks
Change in hemoglobin A1c | 6 weeks
Change in blood pressure | 6 weeks
QT interval | 6 weeks
  Electrocardiograph (ECG) Parameters
PR interval | 6 weeks
  Electrocardiograph (ECG) Parameters
QRS interval | 6 weeks
  Electrocardiograph (ECG) Parameters
Heart Rate | 6 weeks
  Electrocardiograph (ECG) Parameters
Change in body weight | 6 weeks
  Measured by Tanita Body Composition Analyzer
Change in body fat percentage | 6 weeks
  Measured by Tanita Body Composition Analyzer
Change in body water percentage | 6 weeks
  Measured by Tanita Body Composition Analyzer
Change in muscle mass | 6 weeks
  Measured by Tanita Body Composition Analyzer
Change in bone mass | 6 weeks
  Measured by Tanita Body Composition Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Shah, PharmD, Principal Investigator — University of the Pacific
Locations (1):
- Manshadi Heart Institute, Inc., Stockton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Beck RW, Hirsch IB, Laffel L, Tamborlane WV, Bode BW, Buckingham B, Chase P, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Huang ES, Kollman C, Kowalski AJ, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer SA, Wilson DM, Wolpert H, Wysocki T, Xing D. The effect of continuous glucose monitoring in well-controlled type 1 diabetes. Diabetes Care. 2009 Aug;32(8):1378-83. doi: 10.2337/dc09-0108. Epub 2009 May 8. PMID 19429875
- [Background] Food and Drug Administration. Self-monitoring blood glucose test systems for over-the-counter use-guidance for industry and food and drug administration staff. Available at: http://www.fda.gov/downloads/MedicalDevices/DeviceRegulationandGuidance/GuidanceDocuments/UCM380327.pdf. Accessed October 10, 2016.
- [Background] Siegmund T, Heinemann L, Kolassa R, Thomas A. Discrepancies Between Blood Glucose and Interstitial Glucose-Technological Artifacts or Physiology: Implications for Selection of the Appropriate Therapeutic Target. J Diabetes Sci Technol. 2017 Jul;11(4):766-772. doi: 10.1177/1932296817699637. Epub 2017 Mar 21. PMID 28322063
- [Background] Shapiro AR. Nonadjunctive Use of Continuous Glucose Monitors for Insulin Dosing: Is It Safe? J Diabetes Sci Technol. 2017 Jul;11(4):833-838. doi: 10.1177/1932296816688303. Epub 2017 Mar 1. PMID 28540756
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S66-S76. doi: 10.2337/dc20-S006. PMID 31862749
- [Background] Vigersky RA, McMahon C. The Relationship of Hemoglobin A1C to Time-in-Range in Patients with Diabetes. Diabetes Technol Ther. 2019 Feb;21(2):81-85. doi: 10.1089/dia.2018.0310. Epub 2018 Dec 21. PMID 30575414
- [Background] FreeStyle Libre 2-Best Glucose Monitor For Kids - Coming Soon for Patients 4+. Continuous Glucose Monitoring System. https://www.freestylelibre.us/system-overview/freestyle-libre-2.html. Accessed June 21, 2020.
- [Background] Kawatra P, Rajagopalan R. Cinnamon: Mystic powers of a minute ingredient. Pharmacognosy Res. 2015 Jun;7(Suppl 1):S1-6. doi: 10.4103/0974-8490.157990. PMID 26109781
- [Background] Foster M, Hunter D, Samman S. Evaluation of the Nutritional and Metabolic Effects of Aloe vera. In: Benzie IFF, Wachtel-Galor S, editors. Herbal Medicine: Biomolecular and Clinical Aspects. 2nd edition. Boca Raton (FL): CRC Press/Taylor & Francis; 2011. Chapter 3. Available from: https://www.ncbi.nlm.nih.gov/books/NBK92765/